CLINICAL TRIAL: NCT00827359
Title: A Phase II Biomarker Trial of Everolimus in Patients With Advanced Renal Cell Carcinoma
Brief Title: Biomarker Trial of Everolimus in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Duke University (Other); Novartis (Industry)
Responsible Party: Principal Investigator, David F. McDermott, MD, Director of Biologic Therapy Program, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-313
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Renal Cell Carcinoma; Renal Cancer
Keywords: everolimus
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): This is a single-arm study. All patients will receive everolimus.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Tablet form taken orally once a day

SUMMARY:
The purpose of this study is to determine if certain features of tumor specimens sampled prior to therapy can predict for the likelihood of responding to everolimus.

DETAILED DESCRIPTION:
* Participants will undergo a CT or ultrasound guided biopsy of an accessible tumor lesion before beginning the study medication.
* Everolimus tablets will be taken orally once a day. Participants will undergo a physical exam and will be asked questions about their general health and specific questions about any problems they might be having. Photographs will be taken of the tumor to assess the response to treatment. This will be done by a CT or MRI scan. Blood tests will be performed every 4 weeks. In addition, blood for research purposes will be done on day 1 of every other cycle. A urine test will be done every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have at least one site of disease which in the opinion of the investigator is safely accessible by CT guided biopsy or metastasectomy. Safely accessible metastatic disease will be defined to include those lesions which are palpable with no overlying viscera and are at least 2cm in size. Given the paucity of subcutaneous lesions in RCC, lesions which are felt to be safe to biopsy will also be allowed. These lesions include pleural-based tumors, peripheral liver lesions, kidney lesions and bone lesions with exophytic soft tissue component. As with palpable lesions, these other lesions should be at least 2cm in size with no overlying viscera.
* At least one measurable site of disease, other than the biopsy site, according to RECIST criterial that has not been previously irradiated. Th the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Metastatic renal carcinoma with histologic confirmation by the treating center of either primary or a metastatic lesion. Non-clear cell histologies will be allowed
* 18 years of age or older
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
* ECOG Performance status of 1 or less
* Adequate bone marrow, liver and renal function as outlined in the protocol
* Fasting serum cholesterol < 300mg/dL OR < 7.75 mmol/L AND fasting triglycerides < 2.5 x ULN
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Prior treatment with any investigation drug within the preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Treated brain metastases will be allowed. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS: Gamma Knife, LINAC or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection performed within 3 months prio to day 1 will be excluded.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Uncontrolled diabetes mellitus as defined by a fasting serum > 1.5 x ULN
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus
* Patients with active, bleeding diathesis or on systemic anticoagulation. Aspirin is permitted.
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control.
* Patients who have received prior treatment with an mTOR inhibitor.
* Patients with known hypersensitivity to everolimus or other rapamycins or to its excipients.
* History of noncompliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 25
Treated | 24
Completed | 0
Not Completed | 25
Not completed — Progressive Diseas | 19
Not completed — Unacceptable Toxicity | 5
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 64 [52 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — 00- Fully Active
  01- Restricted 02 - Ambulatory and Capable of Self Care
  Participants
    00 | 15
    01 | 9
Prior Lines of Therapy [Median (Full Range); unit: therapies] | 2 [1 to 7]
Histology [Count of Participants; unit: Participants]
  Clear Cell | 18
  Papillary | 4
  Missing | 2
Memorial Sloan Kettering Cancer Center Risk Class [Count of Participants; unit: Participants]
  Favorable (0 risk factors) | 4
  Intermediate (1-2 risk factors) | 14
  High (>=3 risk factors) | 6
International Metastatic Renal-Cell Carcinoma Database Consortium Class [Count of Participants; unit: Participants]
  Favorable (0 risk factors) | 5
  Intermediate (1-2 risk factors) | 19
  High (≥3 risk factors) | 0
Prior Nephrectomy [Count of Participants; unit: Participants]
  Yes, Radical | 21
  Yes, Partial | 1
  No | 0
  Missing | 2
Metastatic Sites [Count of Participants; unit: Participants]
  Bone | 4
  Liver | 8
  Lung | 16
  Brain | 0
  Renal | 6
  Pancreas | 3
  Lymph Nodes, Intra-Abdominal | 11
  Lymph Node, Pulmonary | 7
  Adrenal Glands | 5
  Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Difference in Median Progression Free Survival Time Between Favorable and Unfavorable Biomarker Group
Description: The biomarkers of interest are pS6 and pAkt. Expression will be classified as low, intermediate, or high based on a composite score of staining intensity and % of tumor cells staining positive. The difference in progression free survival (PFS) time in the "low" to "high" groups is analyzed. PFS is the time from start of treatment to disease progression (PD) or death (estimated by Kaplan Meier method)s. Patients without PD and alive are censored at last date patient is known PD-free. PD is defined by Response Evaluation Criteria In Solid Tumors Criteria 1.1 (RECIST) as follows:
  * >20% increase in the sum of the diameters (SD) of target lesions, referencing the smallest SD on study (including baseline). Must be an increase of >5 mm.
  * New lesions or PD of non-target lesions. Must be represent overall disease status change, not a single lesion increase. Patients with PD at the first on-treatment imaging assessment, will remain on study at investigator discretion until later confirmed.
Time Frame: Follow-up time was up to 39 months from treatment start date.
Population: Phospho-Akt and phospho-S6 immunohistochemistry analysis was unsuccessful due to the lack of adequate tissue samples and was not pursued further.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression (PD) or death from any cause as estimated by Kaplan Meier methods. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free. Progression is defined by Response Evaluation Criteria In Solid Tumors Criteria 1.1 (RECIST) as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including baseline if it's the smallest). The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
Time Frame: Follow-up time was up to 39 months from treatment start date.
Population: Twenty-five patients enrolled onto the study between April 2009 and November 2012. One patient became ineligible because of the inability to obtain a pretreatment biopsy sample. A total of 27 tissue samples were successfully obtained from 24 patients, with 3 sets of paired tissues obtained before treatment and while receiving treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 24
months | 3.8 [2.4 to 5.4]

3. Secondary Outcome: Best Overall Response Rate
Description: The best overall response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response recorded on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  CR and PR must meet the following lesion criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
Time Frame: Evaluated while on treatment. Up to 36 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 24
percentage of participants | 4.2 [0.2 to 18.3]

4. Secondary Outcome: Best Overall Response by PI3K-AKT-MTOR Mutation
Description: Next generation sequencing was used to identify participants with PI3K-AKT-MTOR mutations. Best overall response rate was analyzed with mutant versus wild-type pathways. Please see Best Overall Response Rate for response definition.
Time Frame: Evaluated while on treatment. Up to 36 months
Population: Participants were classified as either "mutations" or "no mutations."
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 24
percentage of participants
  Mutation: number analyzed (Participants) | 18
  Mutation | 5.6
  No Mutations: number analyzed (Participants) | 6
  No Mutations | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24)
nausea (Gastrointestinal disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT00827359/Prot_SAP_000.pdf